CLINICAL TRIAL: NCT04510493
Title: Canakinumab in Patients With COVID-19 and Type 2 Diabetes - CanCovDia Trial
Brief Title: Canakinumab in Patients With COVID-19 and Type 2 Diabetes
Acronym: CanCovDia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Novartis (Industry); Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-02008; me20Donath2
Record Dates: First submitted 2020-08-11; First posted 2020-08-12 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Coronavirus Infection; Diabetes Mellitus, Type 2
Keywords: NLRP3; Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2); Coronavirus Disease 19 (COVID-19); IL-1beta; hyperinflammatory syndrome; obesity
MeSH Terms: conditions — Coronavirus Infections; Diabetes Mellitus, Type 2; COVID-19; Obesity | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active treatment arm (Active Comparator): Treatment with Canakinumab i.v. administered over 2 hours
  Interventions: Drug: Canakinumab
- placebo treatment arm (Placebo Comparator): placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canakinumab — Body weight adjusted dose in 250 ml 5% dextrose solution i.v. over 2 hours
  Other Names: Ilaris®
  Arms: active treatment arm
Drug: Placebo — Aqua ad injectabilia in 250 ml 5% dextrose solution i.v. over 2 hours
  Other Names: Aqua ad injectabilia in 250 ml 5% dextrose solution
  Arms: placebo treatment arm

SUMMARY:
The purpose of this study is to evaluate whether Canakinumab has beneficial effects on patients with Type 2 diabetes mellitus and coronavirus disease 19 (COVID19).

DETAILED DESCRIPTION:
Patients with a metabolic syndrome (overweight, diabetes, hypertension) have a particularly bad outcome if infected with severe acute respiratory syndrome coronavirus 2 (SARS-CoV2). This may be explained by an over-activation of the Interleukin-1 (IL-1) beta system. Metabolic stress (increased glucose and lipid levels) induces NOD-, LRR- and pyrin domain-containing protein 3 (NLRP3) -mediated IL-1beta secretion. SARS-CoV2 also activates NLRP3. Therefore, the study proposes that metabolic stress in patients with overweight and diabetes potentiates COVID-19 induced hyperinflammatory syndrome leading to excess mortality in these vulnerable patients. Canakinumab (Ilaris®) is a recombinant, human monoclonal antibody antagonizing IL-1beta by blocking IL-1beta activity. The aim of the study is to investigate the effect of canakinumab in type 2 diabetic patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus
* Body mass index > 25 kg/m² (overweight)
* Hospitalized with COVID-19

Exclusion Criteria:

* Suspected or known untreated active bacterial, fungal, viral, or parasitic infection with the exception of COVID-19
* Treatment with immunomodulators or immunosuppressant drugs, including but not limited to tocilizumab, tumor necrosis factor (TNF) inhibitors and anti-IL-17 agents within 5 half-lives or 30 days (whichever is longer) prior to randomization with the exception of anakinra which is excluded within 5 half-lives only. Note: Immunomodulators (topical or inhaled) for asthma and atopic dermatitis, and corticosteroids (any route of administration) such as dexamethasone are permitted.
* History of hypersensitivity to canakinumab or to biologic drugs
* Neutrophil count <1000/mm3
* Pregnant or nursing (lactating) women
* Participation in another study with investigational drug within the 30 days preceding and during the present study-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
unmatched win ratio after treatment with canakinumab compared to Placebo (composite endpoint) | within 4 weeks after treatment with canakinumab or placebo
  Treatment and placebo will be compared on the basis of the unmatched win-ratio approach of Pocock. When comparing two patients, the winner will be determined by the first component in which the two patients differ (4 weeks after randomization):
  1. longer survival time
  2. longer ventilation-free time
  3. longer ICU-free time
  4. shorter hospitalization time
  If there is no difference between treatment and Placebo: the win ratio is 1. If there is a difference between treatment and Placebo: the win ratio is not 1.

SECONDARY OUTCOMES:
Time to clinical improvement | From randomization up to 4 weeks
  Time to clinical improvement, defined as the time from randomization to either an improvement of two points on a seven-category ordinal scale or discharge from the hospital, whichever comes first. "The seven-category ordinal scale consists of the following categories:
  1. not hospitalized with resumption of normal activities;
  2. not hospitalized, but unable to resume normal activities;
  3. hospitalized, not requiring supplemental oxygen;
  4. hospitalized, requiring supplemental oxygen;
  5. hospitalized, requiring nasal high-flow oxygen therapy, noninvasive mechanical ventilation, or both;
  6. hospitalized, requiring extracorporeal membrane oxygenation (ECMO), invasive mechanical ventilation, or both; and
  7. death"
Death rate | 4 weeks
  Death rate during the 4-week period after study treatment
Admission to intensive care unit (ICU) | 4 weeks
  Admission to the intensive care unit from the medical ward during the 4-week period after study treatment
Secondary worsening of disease | 4 weeks
  Secondary worsening of disease (i.e., development of Acute respiratory distress Syndrome (ARDS), increase of oxygen demand after 72h of treatment)
Prolonged hospital stay | >3 weeks
  Prolonged hospital stay > 3 weeks
Change in ratio to baseline in the glycated hemoglobin | Baseline, Day 29 and Day 90
  Ratio to baseline in the glycated hemoglobin
Change in ratio to baseline in the fasting glucose | Baseline, Day 29
  Ratio to baseline in the fasting glucose
Change in ratio to baseline in the fasting insulin | Baseline, Day 29
  Ratio to baseline in the fasting insulin
Change in ratio to baseline in the fasting c-peptide | Baseline, Day 29
  Ratio to baseline in the fasting c-peptide
Ratio to baseline in the C-reactive protein (CRP) | Baseline, Day 29 and Day 90
  Ratio to baseline in the C-reactive protein (CRP)
Change in ratio to baseline in the D-dimer | Baseline, Day 29
  Ratio to baseline in the D-dimer
Change in ratio to baseline in the Natriuretic peptide (NTproBNP) | Baseline, Day 29 and Day 90
  Ratio to baseline in the Natriuretic peptide (NTproBNP)
Change in ratio to baseline in the Glomerular Filtration Rate Renal (eGFR) | Baseline, Day 29 and Day 90
  Ratio to baseline in the Glomerular Filtration Rate Renal (eGFR)
Type of antidiabetic treatment at Day 29 | Day 29
  Type of antidiabetic treatment at Day 29
Number of antidiabetic treatment at Day 29 | Day 29
  Number of antidiabetic treatment at Day 29
Type of antidiabetic treatment at three months | Month 3
  Type of antidiabetic treatment at three months
Number of antidiabetic treatment at three months | Month 3
  Number of antidiabetic treatment at three months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Donath, MD, Prof., Principal Investigator — University Hospital Basel, Department of Endocrinology, Diabetes and Metabolism
Locations (9):
- Switzerland (9):
  - University Medical Clinic Aarau, Aarau
  - University Hospital Basel, Basel
  - University Hospital Bern, Bern
  - Hopital du Jura, Delémont
  - University Hospital Geneva, Geneva
  - University Hospital Lausanne, Lausanne
  - Cantonal Hospital Lucerne, Lucerne
  - Cantonal Hospital St Gallen, Sankt Gallen
  - University Hospital Zürich, Zurich

REFERENCES:
- [Derived] Hepprich M, Mudry JM, Gregoriano C, Jornayvaz FR, Carballo S, Wojtusciszyn A, Bart PA, Chiche JD, Fischli S, Baumgartner T, Cavelti-Weder C, Braun DL, Gunthard HF, Beuschlein F, Conen A, West E, Isenring E, Zechmann S, Bucklar G, Aubry Y, Dey L, Muller B, Hunziker P, Schutz P, Cattaneo M, Donath MY. Canakinumab in patients with COVID-19 and type 2 diabetes - A multicentre, randomised, double-blind, placebo-controlled trial. EClinicalMedicine. 2022 Sep 17;53:101649. doi: 10.1016/j.eclinm.2022.101649. eCollection 2022 Nov. PMID 36128334